## To whom it may concern:

This is the ethics approval document for the English version of the IIT trial.

Approval Letter of Ethics Committee of National Cancer Center/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College

Approval No.: 19/216-2000 Approval Date: August 15, 2019

**Study Title**: A Real-World Observational Cohort Study on Consolidation Therapy in Patients with Inoperable Locally Advanced Non-Small Cell Lung Cancer Who Have Not Progressed After Thoracic Radiotherapy Combined with Chemotherapy (Protocol No.: NCC-002579)

Protocol No. & Version Date: Version 1.0, Date: 2019-08-08 IC Form Version No. & Date: Version 1.0, Date: 2019-08-08

Drug Name: PD1/PDL1

Clinical Trial Approval No. & Issued by:

Trial Class & Phase: Therapeutic Biopharmaceuticals / Class 1 / Other

Study Site and Principal Investigator: Cancer Hospital, Chinese Academy of Medical Sciences, Bi Nan

Sponsor Name: Cancer Hospital, Chinese Academy of Medical Sciences

## **Evaluation comments:**

The Ethics Committee received your application for new project approval on August 13, 2019, and carefully discussed and voted on the above-mentioned trial protocol, informed consent form and related contents (see attachments) on August 15, 2019. The number of attendees was  $\underline{7}$ , and the number of voters was  $\underline{7}$ . The votes were as follows:  $\underline{3}$  in favor of modification,  $\underline{3}$  in favor of approval after modification,  $\underline{1}$  for re-examination after modification,  $\underline{0}$  against, Termination or suspension of the approved trial:  $\underline{0}$  votes. Approval result: Modified and agreed. The ethics committee suggests further revision of the trial protocol:

The Ethics Committee reviewed the revised trial protocol, informed consent form and IIT ethics application form on June 22, 2020. They considered that the modifications were basically in line with ethical requirements and the clinical research could commence.

The valid time is one year from date of signature of Chairman and extended with annual verification by regulation of Ethics Committee.

Signature of Chairman of the Ethics Committee:

Confidential Date: June 23, 2020

Attachment: List of Files Approved by the Ethics Committee

- 1. Ethical Approval Application Form (Form No. 02)
- 2. List of Study Group Members (Form No. 03)
- 3. CV of the Investigator
- 4. Clinical Trial Protocol (Version No.: 1.0, Version Date: August 8, 2019)
- 5. Ethical Declaration for Investigator-Initiated Study (IIT)
- 6. Informed Consent Form
- 7. Case Report Form Files

Reviewed on June 15, 2020:

1. Trial Protocol (Version No.: 1.1, Version Date: March 28, 2020)

2. Informed Consent Form

3. Ethical Declaration for IIT

4. Revised Abstract

No further text follows

Chairman: 43 2 W

National Cancer Center/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College

National GCP Center for Anticancer Drugs, The Independent Ethics Committee